CLINICAL TRIAL: NCT03619876
Title: Effects of Abatacept on Myocarditis in Rheumatoid Arthritis
Acronym: AMiRA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Laura Geraldino-Pardilla, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS2235
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis; Myocardial Inflammation
Keywords: CTLA4-Ig; Abatacept; Myocarditis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid; Myocarditis | interventions — Abatacept; Adalimumab

STUDY DESIGN:
Intervention Model Description: RA patients will be randomized in an unblinded, 1:1 ratio to treatment with abatacept vs adalimumab. A cardiac FDG PET/CT will be performed at baseline and 16(±2) weeks post-biologic treatment. T cell subpopulations associated with myocardial FDG uptake will be evaluated at both points in time with their transcriptional phenotype outlined by RNAseq.
Masking Description: Unblinded- open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Non- Tumor necrosis factor (TNF) inhibitor arm (Active Comparator): Treatment with abatacept will consist of weekly subcutaneous (SQ) injections at a dose of 125mg.
  Interventions: Drug: Abatacept
- TNF inhibitor arm (Active Comparator): Treatment with a adalimumab, as the TNF-inhibitor arm, will consist of every 2 weeks SQ injections at a dose of 40mg.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Abatacept — 125 MG/ML subcutaneous injections
  Other Names: Orencia
  Arms: Non- Tumor necrosis factor (TNF) inhibitor arm
Drug: Adalimumab — 40 Mg/0.8 mL Subcutaneous Kit
  Other Names: Humira
  Arms: TNF inhibitor arm

SUMMARY:
This study aims to evaluate the effects of abatacept, a CTLA4-Ig fusion protein that binds cluster of differentiation antigen 80 (CD80)/86 (B7-1/B7-2), on subclinical myocarditis in rheumatoid arthritis (RA) through its effect on T cell subpopulations. RA patients without clinical CVD, biologic naïve, and with inadequate response to methotrexate (MTX), will undergo cardiac fluorodeoxyglucose (FDG) positron emission tomography (PET)/computerized tomography (CT) imaging to assess myocardial inflammation. Studies that investigate the impact of treatment on subclinical myocarditis in RA, a possible contributor to heart failure, while exploring potential underlying mechanisms (i.e., different T cell subpopulations), are needed for a better understanding of their relevance in the pathogenesis of heart failure in RA and survival improvement in these patients with excess risk for cardiovascular death. If the investigator hypothesis is confirmed and treatment with abatacept decreases and/or suppresses or prevents myocardial inflammation in RA, this will have multidisciplinary implications that could lead to changes in the current management of RA patients at high risk for cardiovascular events. Similarly, identification of T cell subpopulations in RA patients with myocardial FDG uptake will shed light into the underlying cellular mechanisms of myocardial injury and serve to guide the use of therapies that prevent their pathogenicity. The objectives of this study are to compare the change in myocardial FDG uptake in RA patients treated with abatacept vs adalimumab, and identify T cell subpopulations associated with myocardial FDG uptake in each treatment arm. RA patients will be randomized in an unblinded, 1:1 ratio to treatment with abatacept vs adalimumab. A cardiac FDG PET/CT will be performed at baseline and 16 weeks post-biologic treatment. T cell subpopulations associated with myocardial FDG uptake will be evaluated at both points in time with their transcriptional phenotype outlined by RNA sequencing.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic inflammatory disease that affects ~1% of the population. Regardless of the novel therapies developed in the last decades, studies report an increased standard mortality ratio as high as 3.0 when compared with the general population. Cardiovascular disease (CVD) is the leading cause of mortality in RA subjects in whom the average lifespan is reduced by 8-15 years compared to matched controls. RA patients are at increased risk for developing heart failure and inflammatory myocarditis potentially contributes to this excess risk. Although subclinical myocarditis remains poorly characterized to date in RA, costimulatory molecules such as CD80/86 (B7s) and CD40 are known to play a pivotal role for cytokine production and antigen-specific T cell activation in viral myocarditis, and in murine models, blocking CD40L/B7-1 and CTLA4 significantly decreases myocardial inflammation, damage, and mortality. In addition, the recent increase in the use of immune checkpoint inhibitors for the treatment of numerous cancers, has raised awareness of the occurrence of fulminant autoimmune lymphocytic myocarditis as a complication of these drugs including anti-CTLA4 due to a presumed uncontrolled immune response resulting in T-cell mediated myocardial injury. Interestingly, pilot data showed lower myocardial FDG uptake in RA patients on the a CTLA4-Ig fusion protein abatacept compared with other DMARDs. These data raise the possibility of immunotherapy for the treatment of myocarditis in RA, suggesting a role for T cell infiltration in its pathogenesis, and a particular benefit for treatment with abatacept vs non-abatacept biologic DMARDs.

In a single RHeumatoid arthritis studY of THe Myocardium (RHYTHM study), a total of 119 RA patients without clinical CVD underwent cardiac FDG-PET/CT, with myocardial inflammation assessed qualitatively and quantitatively by visual inspection and by calculation of the standardized-uptake-value (SUV) units. Qualitative myocardial FDG uptake was observed in 39% of the patients. Animal data showing decreased myocardial inflammation, damage, and mortality, and improved cardiac function with CD40L/B7-1 and CTLA4 blockage, coupled with preliminary findings of lower myocardial inflammation in RA patients on abatacept vs other DMARDs, suggest that abatacept treatment has potential myocardial benefits. In RA patients, the proportion of peripheral T cell subsets significantly differs from normal controls and include differentiation to memory effector subsets, acquisition of natural killer (NK) receptors, exhaustion markers, and enhanced inflammatory cytokine expression. Importantly, T cell lymphocytic infiltration described in autoimmune myocarditis resulting as a complication of CTLA4 immune checkpoint inhibition, suggests a role for T cell subsets in the pathogenesis of myocarditis in RA with potential differences depending on mechanism of action of the DMARD in use. Studies that investigate the impact of treatment on subclinical myocarditis in RA, a possible contributor to heart failure, while exploring potential underlying mechanisms (i.e., different T cell subpopulations), are needed for a better understanding of their relevance in the pathogenesis of heart failure in RA and survival improvement in these patients with excess risk for cardiovascular death. If the investigator hypothesis is confirmed and treatment with abatacept decreases and/or suppresses or prevents myocardial inflammation in RA, this will have multidisciplinary implications that could lead to changes in the current management of RA patients at high risk for cardiovascular events. Similarly, identification of T cell subpopulations in RA patients with myocardial FDG uptake will shed light into the underlying cellular mechanisms of myocardial injury and serve to guide the use of therapies that prevent their pathogenicity.

This is a single-center study. Twenty RA patients will be recruited over a planned recruitment period of 24 months, and randomized with aims of enrolling 10 patients per year, the enrollment rate is estimated as 1 patient per month. The target population consists of patients who are deemed methotrexate-inadequate responders by the patient's treating rheumatologist, and who have not yet stepped up to additional treatment with a biologic DMARD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed by the subject.
* Patients age > 18 years.
* Fulfilling the American College of Rheumatology 2010 classification criteria for RA.
* MTX for ≥ 8 weeks at ≥ 15mg weekly or on at least 7.5mg of methotrexate weekly for ≥8 weeks with a documented intolerance of higher MTX doses, and on a stable dose for the previous 4 weeks;
* Naïve to biologic treatment.
* If the subject is a woman with childbearing potential, a urine sample will be taken for a pregnancy test. The results of the pregnancy test must be negative.

Exclusion Criteria:

* Prior biologic use.
* Any prior self-reported physician diagnosed CV event (myocardial infarction; angina; stroke or Transient Ischemic Attack (TIA); heart failure; prior CV procedure (i.e., coronary artery bypass graft, angioplasty, valve replacement, pacemaker).
* Active history of cancer.
* Prior use of immune checkpoint inhibitors.
* Known pregnancy, HIV, hepatitis B, hepatitis C, active (or untreated latent) tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Geraldino-Pardilla, MD, Principal Investigator — CUMC
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Symmons DP, Jones MA, Scott DL, Prior P. Longterm mortality outcome in patients with rheumatoid arthritis: early presenters continue to do well. J Rheumatol. 1998 Jun;25(6):1072-7. PMID 9632066
- [Background] Solomon DH, Karlson EW, Rimm EB, Cannuscio CC, Mandl LA, Manson JE, Stampfer MJ, Curhan GC. Cardiovascular morbidity and mortality in women diagnosed with rheumatoid arthritis. Circulation. 2003 Mar 11;107(9):1303-7. doi: 10.1161/01.cir.0000054612.26458.b2. PMID 12628952
- [Background] Sihvonen S, Korpela M, Laippala P, Mustonen J, Pasternack A. Death rates and causes of death in patients with rheumatoid arthritis: a population-based study. Scand J Rheumatol. 2004;33(4):221-7. doi: 10.1080/03009740410005845. PMID 15370716
- [Background] Solomon DH, Goodson NJ, Katz JN, Weinblatt ME, Avorn J, Setoguchi S, Canning C, Schneeweiss S. Patterns of cardiovascular risk in rheumatoid arthritis. Ann Rheum Dis. 2006 Dec;65(12):1608-12. doi: 10.1136/ard.2005.050377. Epub 2006 Jun 22. PMID 16793844
- [Background] Wolfe F, Freundlich B, Straus WL. Increase in cardiovascular and cerebrovascular disease prevalence in rheumatoid arthritis. J Rheumatol. 2003 Jan;30(1):36-40. PMID 12508387
- [Background] LEBOWITZ WB. The heart in rheumatoid arthritis (rheumatoid disease). A clinical and pathological study of sixty-two cases. Ann Intern Med. 1963 Jan;58:102-23. doi: 10.7326/0003-4819-58-1-102. No abstract available. PMID 13928929
- [Background] CATHCART ES, SPODICK DH. Rheumatoid heart disease. A study of the incidence and nature of cardiac lesions in rheumatoid arthritis. N Engl J Med. 1962 May 10;266:959-64. doi: 10.1056/NEJM196205102661901. No abstract available. PMID 13877345
- [Background] SOKOLOFF L. CARDIAC INVOLVEMENT IN RHEUMATOID ARTHRITIS AND ALLIED DISORDERS: CURRENT CONCEPTS. Mod Concepts Cardiovasc Dis. 1964 Apr;33:847-50. No abstract available. PMID 14144874
- [Background] Han B, Jiang H, Liu Z, Zhang Y, Zhao L, Lu K, Xi J. CTLA4-Ig relieves inflammation in murine models of coxsackievirus B3-induced myocarditis. Can J Cardiol. 2012 Mar-Apr;28(2):239-44. doi: 10.1016/j.cjca.2011.11.014. Epub 2012 Feb 14. PMID 22336520
- [Background] Matsui Y, Inobe M, Okamoto H, Chiba S, Shimizu T, Kitabatake A, Uede T. Blockade of T cell costimulatory signals using adenovirus vectors prevents both the induction and the progression of experimental autoimmune myocarditis. J Mol Cell Cardiol. 2002 Mar;34(3):279-95. doi: 10.1006/jmcc.2001.1511. PMID 11945021
- [Background] Abe S, Hanawa H, Hayashi M, Yoshida T, Komura S, Watanabe R, Lie H, Chang H, Kato K, Kodama M, Maruyama H, Nakazawa M, Miyazaki J, Aizawa Y. Prevention of experimental autoimmune myocarditis by hydrodynamics-based naked plasmid DNA encoding CTLA4-Ig gene delivery. J Card Fail. 2005 Sep;11(7):557-64. doi: 10.1016/j.cardfail.2005.04.005. PMID 16198253
- [Background] Liu W, Gao C, Zhou BG, Li WM. Effects of adenovirus-mediated gene transfer of ICOSIg and CTLA4Ig fusion protein on experimental autoimmune myocarditis. Autoimmunity. 2006 Mar;39(2):83-92. doi: 10.1080/08916930500507870. PMID 16698663
- [Background] Johnson DB, Balko JM, Compton ML, Chalkias S, Gorham J, Xu Y, Hicks M, Puzanov I, Alexander MR, Bloomer TL, Becker JR, Slosky DA, Phillips EJ, Pilkinton MA, Craig-Owens L, Kola N, Plautz G, Reshef DS, Deutsch JS, Deering RP, Olenchock BA, Lichtman AH, Roden DM, Seidman CE, Koralnik IJ, Seidman JG, Hoffman RD, Taube JM, Diaz LA Jr, Anders RA, Sosman JA, Moslehi JJ. Fulminant Myocarditis with Combination Immune Checkpoint Blockade. N Engl J Med. 2016 Nov 3;375(18):1749-1755. doi: 10.1056/NEJMoa1609214. PMID 27806233
- [Background] Varricchi G, Galdiero MR, Tocchetti CG. Cardiac Toxicity of Immune Checkpoint Inhibitors: Cardio-Oncology Meets Immunology. Circulation. 2017 Nov 21;136(21):1989-1992. doi: 10.1161/CIRCULATIONAHA.117.029626. No abstract available. PMID 29158212

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven participants enrolled and 10 randomized. One participant withdrew prior to randomization.
Groups:
- Non-TNF Inhibitor Arm: Treatment with abatacept will consist of weekly subcutaneous (SQ) injections at a dose of 125mg.
  Abatacept: 125 MG/ML subcutaneous injections
Period: Overall Study
Arm/Group | Non-TNF Inhibitor Arm | TNF Inhibitor Arm
Started | 4 | 6
Completed | 3 | 2
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Withdrawal due to incidental finding | 0 | 2

BASELINE CHARACTERISTICS:
Population: Of the four participants that started in the Non-TNF inhibitor arm, three were included in baseline analysis as one participant withdrew. Of the six participants that started in the TNF inhibitor arm, four were included in baseline analysis, as two participants withdrew.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-TNF Inhibitor Arm | TNF Inhibitor Arm | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13.45362) | 44.75 (12.60622) | 50.86 (14.06448)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1
  Hispanic | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Myocardial FDG Uptake in Rheumatoid Arthritis (RA) Patients Treated With Abatacept vs Adalimumab.
Description: Using FDG PET cardiac imaging to identify myocardial inflammation at baseline and post-treatment, the study will quantitatively compare the change in myocardial FDG uptake in biologic naïve RA patients without clinical CVD and with inadequate methotrexate response, following randomization to 16-week treatment with abatacept vs the TNF-inhibitor adalimumab. Conventional cardiovascular disease (CVD) risk factors and measures of RA disease activity and severity will be ascertained.
Time Frame: Baseline, 16 weeks
Population: Zero participants analyzed as none of the participants treated had FDG uptake at any timepoint.
Arm/Group | Non-TNF Inhibitor Arm | TNF Inhibitor Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Prevalence of T Cell Subpopulations Associated With Myocardial FDG Uptake in RA Patients Treated With Abatacept vs Adalimumab.
Description: This is to test whether elevations in different T cell subsets are associated with myocardial FDG uptake in RA patients treated with abatacept vs adalimumab. Subsequently, the transcriptional phenotype of candidate subpopulations.
Time Frame: Baseline, 16 weeks
Population: Zero participants analyzed as none of the participants treated had FDG uptake at any timepoint.
Arm/Group | Non-TNF Inhibitor Arm | TNF Inhibitor Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Non-TNF Inhibitor Arm | TNF Inhibitor Arm
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-TNF Inhibitor Arm (N=3) | TNF Inhibitor Arm (N=2)
Cough (General disorders) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Incidental finding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT03619876/Prot_SAP_000.pdf